CLINICAL TRIAL: NCT01360242
Title: Patients Presenting With Acute STEMI Treated With Primary PCI : Comparison of the Impact of the MIMI Approach With a Conventional Strategy of Immediate Stenting
Brief Title: Minimal Invasive Procedure for Myocardial Infarction
Acronym: MIMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A01345-34
Record Dates: First submitted 2011-04-28; First posted 2011-05-25 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Acute STEMI; Thrombus aspiration; Angioplasty; Primary Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIMI procedure (two-step strategy) (Active Comparator): Thrombus aspiration is performed to achieve TIMI-3 flow. Once TIMI-3 flow is restored and sustained for > 10 minutes, the initial procedure is stopped regardless of the presence of any residual stenosis. A second coronary angiogram is performed 24-48 hours later and the physician is free to decide on the best treatment, i.e. surgery, medical treatment, or stent implantation (drug-eluting stent if indicated for on-label patients). If stenting is required and the thrombus is still too large (greater than twice the artery width), the physician could postpone stent implantation for days or weeks.
  Interventions: Procedure: MIMI procedure (two-step strategy)
- Immediate Stenting (one-step strategy) (Sham Comparator): The physician is encouraged to implant a stent after the thrombus aspiration (drug-eluting stent if indicated for on-label patients).
  Interventions: Procedure: Immediate Stenting (one-step strategy)

INTERVENTIONS:
Procedure: MIMI procedure (two-step strategy) — A second coronary angiogram is performed 24-48 hours later and the physician is free to decide on the best treatment, i.e. surgery, medical treatment, or stent implantation (drug-eluting stent if indicated for on-label patients). If stenting is required and the thrombus is still too large (greater than twice the artery width), the physician could postpone stent implantation for days or weeks.
  Other Names: Delayed angioplasty; Two-step strategy
  Arms: MIMI procedure (two-step strategy)
Procedure: Immediate Stenting (one-step strategy) — The physician is encouraged to implant a stent after the thrombus aspiration (drug-eluting stent if indicated for on-label patients).
  Other Names: Immediate Angioplasty
  Arms: Immediate Stenting (one-step strategy)

SUMMARY:
In the setting of primary Percutaneous Coronary Intervention (PCI), the investigators hypothesize that a 24-48 hour delay strategy of stenting after successful thrombus aspiration and establishment of Thrombolysis In Myocardial Infarction (TIMI)-3 flow with optimal antithrombotic therapy may decrease the risk of MicroVascular Obstruction (MVO) as assessed by Cardiac Magnetic Resonance Imaging (CMRI).

DETAILED DESCRIPTION:
Primary PCI is the reperfusion therapy of choice in patients with acute ST-elevation myocardial infarction (STEMI) [Van de Werf et al. 2008; Kushner et al. 2009]. The first objective in primary PCI is to restore TIMI-3 flow. However, despite restoration of TIMI-3 flow, myocardial reperfusion remains suboptimal in a significant proportion of patients, predominantly as a consequence of the so called "myocardial non-reperfusion phenomenon", "low/no-reflow phenomenon" or MVO. This, in turn, is associated with significant morbidity and mortality [Brodie et al. 2005; Bruder et al. 2008; Hombach et al. 2005; Nijveldt et al. 2008; Thiele et al. 2008; Wu et al. 1998]. Although TIMI flow is well assessed by angiography, contrast-enhanced CMRI remains the gold standard in the assessment of MVO. Indeed, the presence and extent of hypoenhanced areas have been shown to be associated with a poor outcome [Bruder et al. 2008; Hombach et al. 2005; Nijveldt et al. 2008; Wu et al. 1998].

There is now a large body of evidence to suggest that even in patients with TIMI-3 flow on angiography, as many as 60% of these patients will subsequently exhibit MVO with CMRI [Brodie et al. 2005; Bruder et al. 2008; Hombach et al. 2005; Nijveldt et al. 2008; Thiele et al. 2008; Wu et al. 1998]. Our knowledge of the mechanisms of MVO occurrence as well as measures to reduce MVO has been considerably enhanced by recent publications. For instance, Sianos et al. [2007] demonstrated that the thrombus burden at the time of angiography is an independent predictor of MVO extension and 2-year mortality. Furthermore, Isaaz et al. [2006] recommended a two-step strategy as a means of minimising the risk of MVO, with the first step consisting of TIMI-3 flow restoration, followed 2-6 days later by further angiography to determine the therapeutic strategy of choice (PCI, cardiac surgery, or medical treatment: 67%, 25%, and 8% respectively). Meneveau et al. [2009] also adopted a two-step strategy in a small cohort of STEMI patients with TIMI-3 flow and ST-segment regression at the time of the procedure. They demonstrated that a 24-hour delay in stent implantation led to a higher rate of procedural success than immediate stenting. Isaaz et al. [2006] and Meneveau et al. [2009] also reported a decreased thrombus burden and no culprit-artery re-occlusion between the first and the second procedure.

Both the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS) [Svilaas et al. 2008] and the thrombectomy with EXPort catheter in Infarct-Related Artery during primary percutaneous coronary intervention (EXPIRA) [Sardella et al. 2009] studies demonstrated the benefits of thrombus aspiration as the first step in primary PCI prior to either ballooning or direct stenting. However, as the effects of stenting upon MVO in the setting of acute STEMI remain poorly understood, we propose a randomized study to evaluate the benefits of a 24-48-hour delay in stent implantation compared to immediate stenting in patients presenting with acute STEMI who will undergo primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute STEMI presenting within 12 hours of symptom onset, requiring a primary percutaneous coronary intervention; and written informed consent.
* Patients will be randomized during the angiography if the initial TIMI flow is 0 or 1 in a major artery and if TIMI-3 flow can be restored after thrombus aspiration and sustained for 10 minutes.
* Acute STEMI is defined as typical chest pain with 30 minutes of sustained ST-segment elevation >1 mm in two or more consecutive limb leads or >2 mm in two or more precordial leads in the ECG. Major artery is defined as the proximal or mid segment of the left descending artery, the proximal segment of the circumflex artery (before the first marginal), or the right coronary artery before the posterior descendant artery.

Exclusion Criteria:

* Patients less than 18 years' old
* Pregnant and breast feeding women
* Patients with a pacemaker, automated implantable cardioverter-defibrillator (AICD), or left bundle branch block
* Contraindication to abciximab, prasugrel, or clopidogrel
* Cardiac arrest as initial presentation
* Current medical condition with a life expectancy of < 6 months
* Patients not living in France
* Patients in cardiogenic shock
* Culprit artery <2.5 mm
* Absence of informed consent
* Patients with initial TIMI 2 or 3 flow or no TIMI-3 flow restored after thrombus aspiration
* Rescue PCI after fibrinolysis
* Known creatinine clearance < 30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the extent of MVO as assessed by CMRI, expressed as the ratio of MVO/left ventricular mass, in the MIMI and conventional groups. | day of performing CMRI (between the fourth and the seventh day after randomization)
  The primary end-point will be reviewed by an independent CMRI core laboratory blinded to the group and the procedure.
  MVO is defined as a hypoenhanced subendocardial area in the infarction core 2 or 10 minutes after contrast injection (dark zone). The total myocardial infarction is defined as the sum of hypoenhanced (dark zone) and hyperenhanced (white zone) signals 10 minutes after contrast injection. The CMRI procedure will be standardised with a specific documentation.

SECONDARY OUTCOMES:
Comparison of the MIMI approach and the conventional strategy on TIMI flow, myocardial blush, and ST-segment evolution before and after the first procedure. | before and 60-90 minutes after the first procedure
  Measurements: TIMI flow grade and TIMI frame count (a more sophisticated method for measuring the flow) at the end of the procedure; blush (a more precise evaluation than TIMI flow on angiography); and ST-segment evolution on the electrocardiogram (ECG) before and 60-90 minutes after the first procedure (core laboratory).
To measure TIMI flow and myocardial blush at the beginning and at end of the second procedure in the MIMI group, and to compare with those obtained at the end of the first procedure. | at the beginning and one minute after the end of the second procedure
  Measurements: TIMI flow grade, TIMI frame count, and blush at the beginning and at the end of the second procedure.
Thrombus burden assessment, and culprit artery diameter between each procedure in the MIMI group | during each procedure (0-48 hours)
  Measurements: Thrombus volume and artery diameter at the thrombus location during the first and second procedure, and diameter of the implanted stent (done at the core laboratory).
Assessment of the ST-segment after the second procedure in the MIMI group | at the beginning (puncture) and 60-90 min after the end of the second procedure
  Measurements: Maximal ST-segment elevation before and 60-90 minutes after the second procedure (done at the core laboratory).
Assessment of the impact of the MIMI procedure on hospital clinical events, infarction size (on CMRI) and complications due to the second procedure. | from randomisation to an expected average 4 days stay before hospital discharge
  The following hospital critical events and complications that occur after the first procedure will be analyzed: cardiogenic shock, acute pulmonary oedema, recurrent myocardial infarction, culprit artery re-occlusion, stroke, major bleeding [Bovill et al. 1991], evaluation of no flow, coronary dissection, recurrent myocardial infarction, chest pain, decelerating angio flow, recurrent ST elevation, troponin elevation, severe renal insufficiency, access site bleeding, and access artery occlusion.
  Measurement: CMRI infarction size.
Assessment of the clinical impact of the MIMI procedure at 6 months | 6 months after randomization
  Measurements: In both groups, follow-up will be undertaken at 6 months by a phone call to the general practitioner, cardiologist or patient, to report the occurrence of: death, recurrent myocardial infarction, hospitalization(s) for cardiac insufficiency, and unscheduled revascularisation.
Assessment of the microcirculatory resistance in patients in whom a pressure endocoronary wire was used. | after each procedure (0-48 hours)
  Measurement: Index of microcirculatory resistance (IMR) just after stenting (first procedure for the conventional group and second procedure for the MIMI group)
Hospitalization duration for both procedures | expected average time from randomisation to Intensive Care Unit (ICU) discharge of 4 days
  Measurements: Number of days in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Loic BELLE, MD, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (24):
- France (24):
  - CHRA, Annecy
  - Hopital Privé, Antony
  - Ch Bastia, Bastia
  - Clinique Convert, Bourg-en-Bresse
  - CH, Cannes
  - CH, Chambéry
  - CHU, Clermont-Ferrand
  - CHU, Dijon
  - CHU Nord, Grenoble
  - Clinique Mutualiste, Grenoble
  - CHU, Lille
  - CH St Luc St Joseph, Lyon
  - CHU Croix Rousse, Lyon
  - Clinique du Tonkin, Lyon
  - CHU Nord, Marseille
  - CHI, Montfermeil
  - Clinique Marie Lannelongue, Paris
  - CH, Pontoise
  - Clinique de Courlancy, Reims
  - Clinique St Hilaire, Rouen
  - CHU, Saint-Etienne
  - Clinique St Gatien, Tours
  - CH, Valence
  - CH, Vichy

REFERENCES:
- [Background] Bovill EG, Terrin ML, Stump DC, Berke AD, Frederick M, Collen D, Feit F, Gore JM, Hillis LD, Lambrew CT, et al. Hemorrhagic events during therapy with recombinant tissue-type plasminogen activator, heparin, and aspirin for acute myocardial infarction. Results of the Thrombolysis in Myocardial Infarction (TIMI), Phase II Trial. Ann Intern Med. 1991 Aug 15;115(4):256-65. doi: 10.7326/0003-4819-115-4-256. PMID 1906692
- [Background] Brodie BR, Stuckey TD, Hansen C, VerSteeg DS, Muncy DB, Moore S, Gupta N, Downey WE. Relation between electrocardiographic ST-segment resolution and early and late outcomes after primary percutaneous coronary intervention for acute myocardial infarction. Am J Cardiol. 2005 Feb 1;95(3):343-8. doi: 10.1016/j.amjcard.2004.09.031. PMID 15670542
- [Background] Bruder O, Breuckmann F, Jensen C, Jochims M, Naber CK, Barkhausen J, Erbel R, Sabin GV; Herzinfarktverbund Essen. Prognostic impact of contrast-enhanced CMR early after acute ST segment elevation myocardial infarction (STEMI) in a regional STEMI network: results of the "Herzinfarktverbund Essen". Herz. 2008 Mar;33(2):136-42. doi: 10.1007/s00059-008-3102-8. PMID 18344033
- [Background] Hombach V, Grebe O, Merkle N, Waldenmaier S, Hoher M, Kochs M, Wohrle J, Kestler HA. Sequelae of acute myocardial infarction regarding cardiac structure and function and their prognostic significance as assessed by magnetic resonance imaging. Eur Heart J. 2005 Mar;26(6):549-57. doi: 10.1093/eurheartj/ehi147. Epub 2005 Feb 15. PMID 15713695
- [Background] Isaaz K, Robin C, Cerisier A, Lamaud M, Richard L, Da Costa A, Sabry MH, Gerenton C, Blanc JL. A new approach of primary angioplasty for ST-elevation acute myocardial infarction based on minimalist immediate mechanical intervention. Coron Artery Dis. 2006 May;17(3):261-9. doi: 10.1097/00019501-200605000-00010. PMID 16728877
- [Background] Kushner FG, Hand M, Smith SC Jr, King SB 3rd, Anderson JL, Antman EM, Bailey SR, Bates ER, Blankenship JC, Casey DE Jr, Green LA, Hochman JS, Jacobs AK, Krumholz HM, Morrison DA, Ornato JP, Pearle DL, Peterson ED, Sloan MA, Whitlow PL, Williams DO; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2009 Focused Updates: ACC/AHA Guidelines for the Management of Patients With ST-Elevation Myocardial Infarction (updating the 2004 Guideline and 2007 Focused Update) and ACC/AHA/SCAI Guidelines on Percutaneous Coronary Intervention (updating the 2005 Guideline and 2007 Focused Update): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2009 Dec 1;120(22):2271-306. doi: 10.1161/CIRCULATIONAHA.109.192663. Epub 2009 Nov 18. No abstract available. PMID 19923169
- [Background] Meneveau N, Seronde MF, Descotes-Genon V, Dutheil J, Chopard R, Ecarnot F, Briand F, Bernard Y, Schiele F, Bassand JP. Immediate versus delayed angioplasty in infarct-related arteries with TIMI III flow and ST segment recovery: a matched comparison in acute myocardial infarction patients. Clin Res Cardiol. 2009 Apr;98(4):257-64. doi: 10.1007/s00392-009-0756-z. Epub 2009 Feb 9. PMID 19205776
- [Background] Nijveldt R, Beek AM, Hirsch A, Stoel MG, Hofman MB, Umans VA, Algra PR, Twisk JW, van Rossum AC. Functional recovery after acute myocardial infarction: comparison between angiography, electrocardiography, and cardiovascular magnetic resonance measures of microvascular injury. J Am Coll Cardiol. 2008 Jul 15;52(3):181-9. doi: 10.1016/j.jacc.2008.04.006. PMID 18617066
- [Background] Sardella G, Mancone M, Bucciarelli-Ducci C, Agati L, Scardala R, Carbone I, Francone M, Di Roma A, Benedetti G, Conti G, Fedele F. Thrombus aspiration during primary percutaneous coronary intervention improves myocardial reperfusion and reduces infarct size: the EXPIRA (thrombectomy with export catheter in infarct-related artery during primary percutaneous coronary intervention) prospective, randomized trial. J Am Coll Cardiol. 2009 Jan 27;53(4):309-15. doi: 10.1016/j.jacc.2008.10.017. PMID 19161878
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Svilaas T, Vlaar PJ, van der Horst IC, Diercks GF, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Thrombus aspiration during primary percutaneous coronary intervention. N Engl J Med. 2008 Feb 7;358(6):557-67. doi: 10.1056/NEJMoa0706416. PMID 18256391
- [Background] Thiele H, Schindler K, Friedenberger J, Eitel I, Furnau G, Grebe E, Erbs S, Linke A, Mobius-Winkler S, Kivelitz D, Schuler G. Intracoronary compared with intravenous bolus abciximab application in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention: the randomized Leipzig immediate percutaneous coronary intervention abciximab IV versus IC in ST-elevation myocardial infarction trial. Circulation. 2008 Jul 1;118(1):49-57. doi: 10.1161/CIRCULATIONAHA.107.747642. Epub 2008 Jun 16. PMID 18559698
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Wu KC, Zerhouni EA, Judd RM, Lugo-Olivieri CH, Barouch LA, Schulman SP, Blumenthal RS, Lima JA. Prognostic significance of microvascular obstruction by magnetic resonance imaging in patients with acute myocardial infarction. Circulation. 1998 Mar 3;97(8):765-72. doi: 10.1161/01.cir.97.8.765. PMID 9498540
- [Derived] Belle L, Motreff P, Mangin L, Range G, Marcaggi X, Marie A, Ferrier N, Dubreuil O, Zemour G, Souteyrand G, Caussin C, Amabile N, Isaaz K, Dauphin R, Koning R, Robin C, Faurie B, Bonello L, Champin S, Delhaye C, Cuilleret F, Mewton N, Genty C, Viallon M, Bosson JL, Croisille P; MIMI Investigators*. Comparison of Immediate With Delayed Stenting Using the Minimalist Immediate Mechanical Intervention Approach in Acute ST-Segment-Elevation Myocardial Infarction: The MIMI Study. Circ Cardiovasc Interv. 2016 Mar;9(3):e003388. doi: 10.1161/CIRCINTERVENTIONS.115.003388. PMID 26957418